CLINICAL TRIAL: NCT03355365
Title: Autologous, Bone Marrow-Derived Mesenchymal Stem Cell-Derived Neural Progenitor Cells (MSC-NP), Expanded Ex Vivo; Administered Intrathecally
Brief Title: Intrathecal Administration of Autologous Mesenchymal Stem Cell-derived Neural Progenitors (MSC-NP) in Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tisch Multiple Sclerosis Research Center of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TISCHMS-MSCNP-002
Record Dates: First submitted 2017-11-14; First posted 2017-11-28 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Mesenchymal Stem Cells; Neural Progenitors; Autologous; Bone Marrow; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Compassionate crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intrathecal MSC-NP injection (Experimental): Patients will receive six autologous stem cell injections through spinal taps every 2 months over a year.
  Interventions: Biological: Intrathecal MSC-NP injection
- Intrathecal saline injection (Placebo Comparator): Patients will receive six placebo injections through spinal taps every 2 months over a year.
  Interventions: Other: Intrathecal saline injection

INTERVENTIONS:
Biological: Intrathecal MSC-NP injection — MSC-NPs represent a neural subpopulation of MSCs from bone marrow with reduced pluripotency and minimized risk of ectopic differentiation, thus are likely to be more suitable for CNS delivery. Importantly, characterization of MSC-NPs demonstrated their immunoregulatory and trophic properties, and MSC-NPs derived from MS and non-MS patients alike were therapeutically viable.
  Arms: Intrathecal MSC-NP injection
Other: Intrathecal saline injection — Placebo
  Arms: Intrathecal saline injection

SUMMARY:
This is a phase II, double-blinded, placebo-controlled, randomized, cross-over Study designed to determine the efficacy of multiple intrathecal administrations of autologous mesenchymal stem cell-derived neural progenitor cells (MSC-NP) compared to placebo in patients with progressive multiple sclerosis. Efficacy will be measured through assessment of disability outcomes. Study participants will receive six intrathecal injections of culture-expanded autologous MSC-NPs at two month intervals in one year and six lumbar punctures as placebo treatments in a second year.

DETAILED DESCRIPTION:
The IT-MSC-NP treatments and all clinical assessments will take place at a single center (Tisch MSRCNY). Study subjects will be assigned to blocks stratified by baseline EDSS score (3.0-4.0, 4.5-5.5, 6.0, and 6.5) and disease subtype (SPMS or PPMS). Study subjects are randomized in an equal fashion (1:1) to study treatment and placebo at initial randomization. Subjects in each block will be randomized into placebo or treatment group. In the second year, treated subjects will cross over to the placebo group and placebo subjects will cross over to the treated group.

The total study duration will be 3 years upon enrollment. Each study subject will be required to attend up to 18 study visits, to include 1 screening visit, 1 bone marrow visit, 1 baseline visit, followed by study visits every 2 months during the treatment period of two years (12 treatment/LP procedure visits and 2 outcome visits), and an additional follow-up visit at the end of year 3.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS as defined by the McDonald criteria
* Diagnosis of primary progressive or secondary progressive MS
* Between the ages of 18-65 years
* Significant disability shown by an Expanded Disability Status Score (EDSS) of greater than or equal to 3.0, and less than or equal to 6.5, that was not acquired within the last 12 months.
* Stable disease state as evidenced by a lack of gadolinium-enhancing lesions on an MRI and by a stable MRI disease burden (number of T2 lesions and size of lesions) in the last six months and no significant change in EDSS (1 point or more) in the last 12 months
* Must agree to undergo four MRIs: at the time of enrollment, after year 1, after year 2, and after year 3
* Patients either within the geographical area or who are able to arrange reliable travel during the study period

Exclusion Criteria:

* EDSS greater than 6.5
* Duration of Disease >20 years at time of screening
* Change of disease modifying agent < 12 months prior to beginning treatment. Additionally, no changes in disease modifying agent will be made during the course of the study.
* Change in MS symptom management treatment < 6 months prior to beginning treatment. Additionally, no changes in MS symptom management treatments will be made during the course of the study, unless there has been clinical improvement, in which case, a patient may discontinue a medication.
* Start of any new orthotic device or durable medical equipment < 6 months prior to beginning treatment or during the course of the study (patients may discontinue use of these devices during the course of the study if they show clinical improvement).
* All patients who have ever been on Lemtrada (alemtuzumab)
* All patients who have had any prior stem cell treatments, including HSCT
* Pregnant or nursing mothers, or any woman intending to become pregnant in the next three years
* All patients will have screening blood tests done. Only patients whose values are in the normal range as determined by the laboratory norms based on age and sex will be allowed to participate. Exceptions may be made for borderline normal laboratory values manifesting no clinical symptoms at the discretion of the Principal Investigator.
* Use of systemic chemotherapeutic or anti-mitotic medications within three months of study start date due to the possibility of interference with bone marrow procedure
* Any patients with a history of or with active malignancy
* Use of steroids within three months of the study start date, as this would suggest an active disease state
* History of cirrhosis due to increased risk of central nervous system (CNS) infection
* Significantly uncontrolled hypertension because of increased risk for stroke or CNS hemorrhage.
* Patients with active thyroid disease resulting in hyperthyroidism or hypothyroidism (Only well controlled patients with labs in the normal range will be included) because of hormone influence on cell growth
* History of central nervous system infection or immunodeficiency syndromes due to increased risk of CNS infection
* Preexisting blood disease (such as bone marrow hypoplasia, leukopenia, thrombocytopenia, or significant anemia) due to invasive nature of bone-marrow aspiration
* Previous or current history of a coagulation disorder
* Any metal implant in the body, which is contraindicated for MRI studies
* Patients with alcohol or other substance abuse problems that may affect stem cell growth; habitual drug (including marijuana and nicotine) abusers, will be excluded from the study
* Other major disease that, in the opinion of the Principal Investigator, would preclude participation in the study
* Patients with Hepatitis B (HBV), Hepatitis C (HCV), syphilis, HIV-1, or HIV-2.
* Any evidence of significant cognitive dysfunction based on a screening history and physical examination because it would preclude giving a truly informed consent
* Patients who are enrolled in another clinical trial for MS treatment or who have received any study drug/biologics within the last 6 months. Additionally, while in the trial, patients may not enroll in any other clinical trial for MS or any other condition.
* Patients who are anticipated to have difficultly accessing the intrathecal space related to scoliosis, obesity, or any other relevant factors determined by the PI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saud A Sadiq, MD, FAAN, Principal Investigator — Tisch MS Research Center of New York
Locations (1):
- Tisch MS Research Center of New York, New York, New York, United States

REFERENCES:
- [Background] Harris VK, Stark J, Vyshkina T, Blackshear L, Joo G, Stefanova V, Sara G, Sadiq SA. Phase I Trial of Intrathecal Mesenchymal Stem Cell-derived Neural Progenitors in Progressive Multiple Sclerosis. EBioMedicine. 2018 Mar;29:23-30. doi: 10.1016/j.ebiom.2018.02.002. Epub 2018 Feb 3. PMID 29449193
- [Result] Harris VK, Stark J, Williams A, Roche M, Malin M, Kumar A, Carlson AL, Kizilbash C, Wollowitz J, Andy C, Gerber LM, Sadiq SA. Efficacy of intrathecal mesenchymal stem cell-neural progenitor therapy in progressive MS: results from a phase II, randomized, placebo-controlled clinical trial. Stem Cell Res Ther. 2024 May 23;15(1):151. doi: 10.1186/s13287-024-03765-6. PMID 38783390

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment First, Then Placebo: Participants will receive six autologous stem cell injections through spinal taps every 2 months over a year. After a period of 3 months, participants will crossover into the placebo group and receive six intrathecal injections of saline every 2 months over a year.
- Placebo First, Then Treatment: Participants will receive six placebo injections through spinal taps every 2 months over a year. After a period of 3 months, participants will crossover into the treatment group and receive six autologous stem cell injections every 2 months over a year.
Period: Year 1, First Intervention
Arm/Group | Treatment First, Then Placebo | Placebo First, Then Treatment
Started | 27 | 27
Completed | 24 | 27
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — pandemic travel limitation | 1 | 0
Period: Year 2, Crossover Intervention
Arm/Group | Treatment First, Then Placebo | Placebo First, Then Treatment
Started | 24 | 27
Completed | 22 | 25
Not Completed | 2 | 2
Not completed — pandemic travel limitation | 1 | 0
Not completed — Adverse event as a result of long-COVID | 1 | 0
Not completed — severe COVID | 0 | 1
Not completed — failure to isolate MSCs from bone marrow | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment First, Then Placebo: Participants will receive six intrathecal injections of autologous stem cells every 2 months over a year. After a 3 month pause, participants will crossover into the placebo group and receive six intrathecal injections of saline every 2 months over a year.
- Placebo First, Then Treatment: Participants will receive six intrathecal injections of saline every 2 months over a year. After a 3 month pause, participants will crossover into the treatment group and receive six intrathecal injections of autologous stem cells every 2 months over a year.
- Total: Total of all reporting groups
Arm/Group | Treatment First, Then Placebo | Placebo First, Then Treatment | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (7) | 49 (9) | 50 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 9 | 7 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline EDSS (expanded disability status scale) [Count of Participants; unit: Participants] — The Expanded Disability Status Scale (EDSS) is a standardized measure used to assess and track the level of disability in people with multiple sclerosis (MS), ranging from 0 (normal neurological status) to 10 (death due to MS) in 0.5 increments. Only ambulatory subjects were enrolled in this study with an EDSS between 3.0 and 6.5. Subgroups of participants were analyzed based on the degree of walking disability. EDSS 3.0-5.5 represents moderate to severe disability but able to walk without assistance, and EDSS 6.0-6.5 represents a need for unilateral or bilateral assistance to ambulate.
  Participants
    EDSS 3.0-5.5 | 14 | 14 | 28
    EDSS 6.0-6.5 | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Expanded Disability Status Scale (EDSS) Plus
Description: Changes in disability assessed based on composite score of EDSS, timed 25-foot walk (T25FW), and nine hole peg test (9HPT) (EDSS-Plus). Improvement is defined by at least one of the following three measures: ≥0.5 decrease in EDSS (if EDSS at entry is ≥ 6.0) or ≥ 1.0 decrease in EDSS (if EDSS at entry is ≤5.5), ≥20% increase in T25FW, or ≥20% increase in 9HPT in either dominant or non-dominant hand. Assessments were made at baseline and month 13. The number of patients who improved in any of the 3 composite measures in month 13 compared to baseline is reported.
Time Frame: Baseline and 13 months
Population: There is no washout period after stem cell injections, therefore outcome measures in participants receiving placebo second in the sequence (treatment first, then placebo) may reflect sustained effects of stem cell treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (IT MSC-NP): Participants received six intrathecal injections of autologous stem cells every 2 months over a year. Assessments were made 3 months after the last injection and compared to baseline. As part of the crossover study, participants were treated either first in the sequence (treatment first, then placebo) or second in the sequence (placebo first, then treatment).
- Placebo (IT Saline): Participants received six intrathecal injections of saline every 2 months over a year. Assessments were made 3 months after the last injection and compared to baseline. As part of the crossover study, participants received placebo either first in the sequence (placebo first, then treatment) or second in the sequence (treatment first, then placebo).
Arm/Group | Treatment (IT MSC-NP) | Placebo (IT Saline)
Number analyzed (Participants) | 49 | 49
Participants | 17 | 17
Statistical Analysis 1: Comparison: Treatment (IT MSC-NP) vs Placebo (IT Saline); Test type: Superiority; p = 1.0, Fisher Exact

2. Secondary Outcome: Change in Multiple Sclerosis Functional Composite (MSFC) Z-Score From Baseline
Description: The Multiple Sclerosis Functional Composite (MSFC) is a standardized tool used to quantify disability in people with multiple sclerosis (MS) by measuring leg function/ambulation (timed 25 foot walk), arm/hand function (9-hole peg test), and cognitive function (Paced Auditory Serial Addition Test). Each assessment is converted into a Z score. A Z-score of 0 represents the population mean. The composite MSFC Z-score represents an average of the 3 Z-scores. A positive change in composite Z-score in month 13 compared to baseline represents better performance and a negative change in composite Z score indicates worse performance.
Time Frame: Baseline and 13 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in composite z score
Arm/Group | Treatment (IT MSC-NP) | Placebo (IT Saline)
Number analyzed (Participants) | 49 | 49
change in composite z score | -.13 (0.85) | -.06 (0.3)
Statistical Analysis 1: Comparison: Treatment (IT MSC-NP) vs Placebo (IT Saline); Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in EDSS From Baseline
Description: The Expanded Disability Status Scale (EDSS) is a standardized measure used to assess and track the level of disability in people with multiple sclerosis (MS), ranging from 0 (normal neurological status) to 10 (death due to MS) in 0.5 increments. Only ambulatory subjects were enrolled in this study with an EDSS between 3.0 and 6.5. Subgroups of participants were analyzed based on the degree of walking disability. EDSS 3.0-5.5 represents moderate to severe disability but able to walk without assistance, and EDSS 6.0-6.5 represents a need for unilateral or bilateral assistance to ambulate. A decrease in EDSS at month 13 compared to baseline is considered improvement.
Time Frame: Baseline and 13 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Treatment (IT MSC-NP) | Placebo (IT Saline)
Number analyzed (Participants) | 49 | 49
change in score on a scale | -0.12 (0.67) | -0.15 (0.77)
Statistical Analysis 1: Comparison: Treatment (IT MSC-NP) vs Placebo (IT Saline); Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percent Change in T25FW (Timed 25 Foot Walk) From Baseline
Description: The timed 25-foot walk (T25FW) is a test used in multiple sclerosis (MS) to assess a person's mobility and leg function, where individuals walk 25 feet as quickly and safely as possible, and the time taken is recorded. A positive percentage change indicates improved walking in month 13 compared to baseline, whereas a negative percentage change indicates worsening.
Time Frame: Baseline and 13 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Treatment (IT MSC-NP) | Placebo (IT Saline)
Number analyzed (Participants) | 49 | 49
% change | -14.4 (41.1) | -19.8 (49.2)
Statistical Analysis 1: Comparison: Treatment (IT MSC-NP) vs Placebo (IT Saline); Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percent Change in 6MWT (6 Minute Walk Test) From Baseline
Description: The 6-minute walk test (6MWT) in multiple sclerosis (MS) measures functional walking capacity by assessing the distance a person can walk in 6 minutes. A positive percentage change indicates improved walking capacity at month 13 compared to baseline, whereas a negative percentage change indicates worsening.
Time Frame: Baseline and 13 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Treatment (IT MSC-NP) | Placebo (IT Saline)
Number analyzed (Participants) | 49 | 49
% change | -15.9 (33.9) | -13.5 (29.7)
Statistical Analysis 1: Comparison: Treatment (IT MSC-NP) vs Placebo (IT Saline); Test type: Superiority; p = .43, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percent Change in 9HPT-D (9 Hole Peg Test in Dominant Hand) From Baseline
Description: The Nine-Hole Peg Test (9HPT) is a standardized, quantitative assessment used to measure manual dexterity and upper extremity function in individuals with multiple sclerosis (MS). Each hand, dominant (D) and non-dominant (ND) is assessed seperately. A positive percentage change indicates improved function at month 13 compared to baseline, whereas a negative percentage change indicates worsening.
Time Frame: Baseline and 13 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Treatment (IT MSC-NP) | Placebo (IT Saline)
Number analyzed (Participants) | 49 | 49
% change | -2.1 (18.1) | -2.9 (17.9)
Statistical Analysis 1: Comparison: Treatment (IT MSC-NP) vs Placebo (IT Saline); Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percent Change in 9HPT-ND (9 Hole Peg Test in Non-Dominant Hand) From Baseline
Description: as for outcome 6
Time Frame: Baseline and 13 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Treatment (IT MSC-NP) | Placebo (IT Saline)
Number analyzed (Participants) | 49 | 49
% change | -4.4 (30.0) | -4.1 (15.0)
Statistical Analysis 1: Comparison: Treatment (IT MSC-NP) vs Placebo (IT Saline); Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in MSWS-12 (12 Item MS Walking Scale) Score From Baseline
Description: The 12-item Multiple Sclerosis Walking Scale (MSWS-12) is a patient-reported outcome measure that assesses the impact of multiple sclerosis (MS) on walking ability. The self-administered questionnaire consists of 12 items addressing how MS has affected various aspects of walking over the past two weeks. Each of the 12 items is scored from 1 to 5 from: 1 = Not at all to 5 = Extremely. Raw total score ranges from 12 (no impairment) to 60 (maximum impairment). Raw score is converted to a standardized score (0-100 scale) producing a final score from 0 = No impact of MS on walking to 100 = Maximum impact. The change in score from baseline to post-intervention was calculated. A decrease in score at month 13 compared to baseline was considered improvement.
Time Frame: Baseline and 13 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in score
Arm/Group | Treatment (IT MSC-NP) | Placebo (IT Saline)
Number analyzed (Participants) | 49 | 49
change in score | -.15 (12.2) | -.15 (15.1)
Statistical Analysis 1: Comparison: Treatment (IT MSC-NP) vs Placebo (IT Saline); Test type: Superiority; p = .71, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in PASAT (Paced Auditory Serial Addition Test) Score From Baseline
Description: The Paced Auditory Serial Addition Test (PASAT) is a neuropsychological test used to assess cognitive impairments, attention, information processing speed, and working memory. The test involves listening to a series of single-digit numbers and the individual must add each new number to the one immediately before it. The score is the number of correct responses out of 60 items. The change in score from baseline to post-intervention is calculated. A positive change in score means an increase in the number of correct answers at month 13 compared to baseline, generally indicating improvement in information processing speed and sustained attention.
Time Frame: Baseline and 13 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in score
Arm/Group | Treatment (IT MSC-NP) | Placebo (IT Saline)
Number analyzed (Participants) | 49 | 49
change in score | 2.3 (5.5) | 1.4 (8.2)
Statistical Analysis 1: Comparison: Treatment (IT MSC-NP) vs Placebo (IT Saline); Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were documented in the intent-to-treat population for the duration of the 2 year study. Year 1 included the MSC-NP group year 1, and the saline group year 1. Study year 2 completed the compassionate crossover design, where subjects treated with saline in year 1 were treated with MSC-NP in year 2, and subjects treated with MSC-NP in year 1 received saline in year 2.
Groups:
- Intrathecal MSC-NP Injection (Year 1): Patients will receive six autologous stem cell injections through spinal taps every 2 months in year 1.
- Intrathecal Saline Injection (Year 1): Patients will receive six placebo injections through spinal taps every 2 months in year 1.
  Intrathecal saline injection: Placebo
- Intrathecal MSC-NP Injection (Year 2): Compassionate crossover design with subjects who were treated with saline/placebo in year 1 received MSC-NP injections in year 2.
- Intrathecal Saline Injection (Year 2): Compassionate crossover design with subjects who were treated with MSC-NP in year 1 received saline injections in year 2.
Arm/Group | Intrathecal MSC-NP Injection (Year 1) | Intrathecal Saline Injection (Year 1) | Intrathecal MSC-NP Injection (Year 2) | Intrathecal Saline Injection (Year 2)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/27 | 0/27 | 3/27 | 3/24
Other Adverse Events (participants affected / at risk) | 24/27 | 15/27 | 20/27 | 13/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intrathecal MSC-NP Injection (Year 1) (N=27) | Intrathecal Saline Injection (Year 1) (N=27) | Intrathecal MSC-NP Injection (Year 2) (N=27) | Intrathecal Saline Injection (Year 2) (N=24)
infection (Infections and infestations) | 1 | 0 | 0 | 0 — Severe urinary tract infection and urosepsis requiring hospitalization.
hyperparathyroid (Endocrine disorders) | 1 | 0 | 0 | 0 — Previously undiagnosed hyperparathyroidism requiring parathyroidectomy. Chronic hypercalcemia contributed to urinary tract infection and sepsis.
infection (Infections and infestations) | 0 | 0 | 1 | 0 — Lung infection associated with long COVID
infection (Infections and infestations) | 0 | 0 | 1 | 0 — Acute appendicitis complicated by bowel perforation.
Muscle weakness (Nervous system disorders) | 0 | 0 | 1 | 0 — Bilateral muscle weakness associated with MS progression
pulmonary embolism (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — Pulmonary embolism and deep vein thrombosis associated with long COVID
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 — COVID-19 infection and severe urinary tract infection
Cholecystitis (Infections and infestations) | 0 | 0 | 0 | 1 — Cholecystitis requiring cholecystectomy
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intrathecal MSC-NP Injection (Year 1) (N=27) | Intrathecal Saline Injection (Year 1) (N=27) | Intrathecal MSC-NP Injection (Year 2) (N=27) | Intrathecal Saline Injection (Year 2) (N=24)
Urinary tract infection (Infections and infestations) | 4 | 3 | 3 | 2
upper respiratory infection (Infections and infestations) | 1 | 2 | 6 | 5
back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
generalized muscle weakness (Nervous system disorders) | 2 | 4 | 2 | 1
Muscle weakness lower limb (Nervous system disorders) | 2 | 1 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 2 | 1 | 1 | 0
Graft vs host disease (Infections and infestations) | 0 | 0 | 1 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
allergic reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
fever (General disorders) | 1 | 0 | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
neck. pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
neuralgia (Nervous system disorders) | 2 | 1 | 0 | 0
paresthesia (Nervous system disorders) | 2 | 0 | 0 | 0
skin infection (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
spasticity (Nervous system disorders) | 1 | 0 | 0 | 1
trigeminal nerve disorder (Nervous system disorders) | 1 | 0 | 1 | 0
vertigo (General disorders) | 1 | 0 | 0 | 1
Headache (General disorders) | 18 | 13 | 18 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT03355365/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT03355365/SAP_001.pdf
  • Informed Consent Form (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT03355365/ICF_002.pdf